CLINICAL TRIAL: NCT03811990
Title: Does a Phone-based Meditation Application Improve Mental Wellness in Emergency Medicine Personnel?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-04-0089
Record Dates: First submitted 2019-01-16; First posted 2019-01-22 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Burnout, Professional; Depression; Anxiety; Stress
MeSH Terms: conditions — Burnout, Professional; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, non-blinded, control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Active Comparator)
  Interventions: Behavioral: Cleveland Clinic Stress Free Now Meditations For Healers

INTERVENTIONS:
Behavioral: Cleveland Clinic Stress Free Now Meditations For Healers — Phone-based meditation application
  Arms: Intervention

SUMMARY:
Emergency medicine is notorious for its high rate of burnout and mental health issues. The emergency department (ED) is a high paced work environment dealing with life and death issues. Employees in the ED work shift times that are not conducive to a natural circadian rhythm. All of these factors lead to high rates of burnout and overall dissatisfaction with their career choice. These are known downsides of a career in emergency medicine, but little effort is put into addressing this issue in everyday EDs.

Cell phones offer an easy and convenient means to participate in meditation. There are multiple evidence-based meditation apps available to cell phone users free of charge. Meditation has been shown to decrease burnout, rates of depression, and rates of anxiety. We hypothesize that weekly use of a meditation-based cell phone application will improve the mental health of emergency department employees as measured on various wellness inventories.

ELIGIBILITY:
Inclusion Criteria:

* Employment in the Emergency Department (with at least 8 shifts a month at Dell Seton Medical Center or Seton Medical Center) as either an attending physician, resident physician, or nurse
* Age greater than/equal to 18 years old and younger than 75 years old
* Must own a mobile phone operating on the iOS system

Exclusion Criteria:

* Already use a phone-based meditation app on a weekly basis
* Currently undergoing psychological treatment in the form of weekly therapy or psychotropic medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in depression score | 90 and 180 days
  Beck Depression Inventory, numeric score of 0-63 with a score of 63 being the most depressed
Change in anxiety score | 90 and 180 days
  Beck Anxiety Inventory, numeric score of 0-63 with a score of 63 being the most anxious
Change in stress levels | 90 and 180 days
  Perceived Stress Scale, numeric score of 0-40 with a score of 40 being the most stressed
Change in burnout level | 90 and 180 days, numeric scale between 0 and 6 with 6 being the highest score
  Maslach Burnout Inventory, measures level of stress on a numeric scale

CONTACTS AND LOCATIONS:
Overall Officials: Keith Lambert, MD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coulon SM, Monroe CM, West DS. A Systematic, Multi-domain Review of Mobile Smartphone Apps for Evidence-Based Stress Management. Am J Prev Med. 2016 Jul;51(1):95-105. doi: 10.1016/j.amepre.2016.01.026. Epub 2016 Mar 15. PMID 26993534